CLINICAL TRIAL: NCT02037360
Title: Mobile Mindfulness Training for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Judson Brewer, Director of Research, Center for Mindfulness, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1305012015
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Smoking Cessation
Keywords: Smoking; Cessation
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Comparator App/Training (Active Comparator): This is a standard smoking cessation smartphone app using the latest evidence-based smoking cessation methods and behavior change theory. Subjects will be encouraged to set a quit date of 3 weeks, to allow comparison to experimental arm quit date.
  Interventions: Behavioral: Active Comparator App/Training
- Experimental App/Training (Experimental): This is a 3-week smartphone-based training program that trains mindfulness for smoking cessation by helping smokers self-monitor their smoking habits, recognize when and how often they smoke, identify triggers for smoking, and learn methods to become more mindful of triggers, to quit smoking with a target quit date of 3 weeks.
  Interventions: Behavioral: Experimental App/Training

INTERVENTIONS:
Behavioral: Active Comparator App/Training — This is a free smoking cessation smartphone app using the latest evidence-based smoking cessation methods and behavior change theory. The app allows users to set a quit date, financial goals, and reminders, track daily smoking habits with an easy-to-use calendar, see graphs tracking money saved and number of packs not smoked, receive health milestones and craving tips to stay motivated, connect with social networks to give milestone updates, create a video diary, and watch personalized video messages from loved ones
  Arms: Active Comparator App/Training
Behavioral: Experimental App/Training — It is comprised of twenty-two modules of 10-15 minutes each, designed to teach mindfulness for smoking cessation using psychoeducation-based audio and videos, animations to reinforce key concepts, and in vivo exercises. In addition, 5 bonus modules become available upon completion of earlier modules; these may be accessed for additional practices to bolster other modules.
  Arms: Experimental App/Training

SUMMARY:
The purpose of this study is to assess the effectiveness of a Mobile Mindfulness Training smartphone application on smoking cessation in smokers ages 18 to 65 years.

DETAILED DESCRIPTION:
In this study, a pilot phase will be carried out first to test feasibility and engagement of the tested intervention. Then in the randomized control trial, subjects will be randomly assigned to receive one of two treatments: (1) a standard smartphone application to support smokers working to become quit-free, or (2) the tested intervention, an app that trains mindfulness for smoking cessation. The primary endpoint of interest will be 1-week point prevalence abstinence at end of treatment, and at 3 and 6 months follow-up for individuals.

ELIGIBILITY:
Inclusion Criteria:

Participants must be (a) 18-65 years of age; (b) smoke 5+ cigarettes/day, (c) < 3 months abstinence in the past year; (d) have a smartphone; and motivated to quit smoking.

Exclusion Criteria:

There are no exclusion criteria. We aim to recruit a heterogeneous group, representative of the general population.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1251 (Actual)
Dates: Start 2015-08; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Point prevalence abstinence at 6 months | 6 months after beginning treatment
  Subjects will be assessed for smoking abstinence at a 6-month follow-up.

SECONDARY OUTCOMES:
Point prevalence abstinence at 3 months | 3 months after beginning treatment
  Subjects will be assessed for smoking abstinence at a 3-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Judson Brewer, MD PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts, Worcester, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Jackson S, Brown J, Norris E, Livingstone-Banks J, Hayes E, Lindson N. Mindfulness for smoking cessation. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD013696. doi: 10.1002/14651858.CD013696.pub2. PMID 35420700
- See also: Click here for more information and to sign up for the study — http://www.umassmed.edu/cfm/Research/Participate-in-Study/